CLINICAL TRIAL: NCT07227415
Title: AN INTERVENTIONAL PHASE 1B/2 STUDY TO EVALUATE THE SAFETY AND EFFICACY OF PF-08634404 MONOTHERAPY AND IN COMBINATION WITH OTHER ANTICANCER AGENTS IN ADULT PARTICIPANTS WITH LOCALLY ADVANCED OR METASTATIC RENAL CELL CARCINOMA
Brief Title: A Study to Learn About the Medicine Called PF-08634404 Dosed Alone and in Combination With Other Anticancer Therapies in Adults With Locally Advanced or Metastatic Renal Cell Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C6461008; 2025-523524-53-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Renal Cell; Advanced Renal Cell Carcinoma; Renal Cancer; Renal Neoplasm; Clear Cell Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Clear-cell Metastatic Renal Cell Carcinoma; Carcinoma, Renal Cell Metastasis; Advanced or Metastatic Renal Cell Carcinoma; Carcinoma, Renal Cell, Advanced; Metastatic Renal Cell Cancer; Metastatic Renal Cell Carcinoma ( mRCC); Metastatic/Advanced Renal Cell Carcinoma
Keywords: Renal cell carcinoma; renal cancer; renal neoplasm
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Clear-cell metastatic renal cell carcinoma; Carcinoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (Experimental): Participants will receive PF-08634404 IV.
  Interventions: Biological: PF-08634404
- Cohort B (Experimental): Participants will receive PF-08634404 in combination with drug 1.
  Interventions: Biological: PF-08634404; Drug: Combination 1
- Cohort C (Experimental): Participants will receive PF-08634404 IV in combination with drug 2.
  Interventions: Biological: PF-08634404; Drug: Combination 2

INTERVENTIONS:
Biological: PF-08634404 — Concentrate for solution for infusion
  Other Names: SSGJ-707
Drug: Combination 1 — Combination Drug 1
  Arms: Cohort B
Drug: Combination 2 — Combination Drug 2
  Arms: Cohort C

SUMMARY:
This study is testing a new medicine called PF-08634404 and how it works in adults with advanced Renal Cell Carcinoma (RCC)- a type of kidney cancer that is either locally advanced (spread to nearby tissues) or metastatic (spread to other parts of the body). The study will look at the safety of the study medicine, when given alone or with other anticancer medicines, and how this type of cancer responds to them.

To join the study, participants must be adults; with locally advanced or metastatic RCC; who have not received treatment for their advanced kidney cancer.

Participants will receive study medicine either alone or with other anticancer medicines. The medicine will be given through intravenous (IV) infusions, which means it will be injected directly into a vein. All treatments will take place at clinical study sites, where trained medical staff will take care of participants during and after each visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at screening
* Locally advanced (not amenable to curative surgery or radiation therapy) or metastatic RCC with diagnosis confirmed by histology/cytology
* At least one measurable (as defined by the investigator) and untreated lesion
* Adequate hematologic, hepatic, cardiac and renal function
* No prior systemic therapy for RCC (immunotherapy after surgery is allowed if received >12 months prior)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* All International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) based risk categories.

Exclusion Criteria:

Participants may be excluded if they meet any of the following:

* Known active brain lesions including leptomeningeal metastasis, brainstem, meningeal or spinal cord metastases or compression.
* Clinically significant risk of haemorrhage or fistula
* History of another malignancy within 3 years
* History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* active autoimmune diseases requiring systemic treatment within the past 2 years
* uncontrolled cardiac and other comorbidities within 6 months prior to the first dose
* Major surgery or severe trauma within 4 weeks before the first dose, or planned major surgery during the study
* History of severe bleeding tendency or coagulation dysfunction
* History of oesophageal varices, severe ulcers, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess
* Acute, chronic or symptomatic infections
* Participants with history of immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-12-04 (Estimated); Primary Completion 2027-11-02 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Confirmed objective response rate (ORR) using RECIST v1.1 as assessed by investigator | Up to approximately 3 years
  ORR is defined as the proportion of participants in the analysis population having a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST v1.1 as assessed by investigator.
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through 90 days after the last study intervention (Up to approximately 3 years)
  AEs as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study intervention.
Number of participants with dose limiting toxicity (DLT) | Though end of DLT evaluation period (Up to approximately 3 years)
  The number of participants who experienced DLTs during the DLT evaluation period in Cohort B (combination 1) and Cohort C (combination 2).

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST v1.1 by investigator | Up to approximately 3 years
  DOR is defined as the time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of first documented disease progression per RECIST v1.1 or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) per RECIST v1.1 by investigator | Up to approximately 3 years
  Progression-free survival is defined as the time from the date of randomization to the date of the first documentation of objective progressive disease (PD) assessed by investigator per RECIST v1.1, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 3 years
  Overall survival defined as the time from the date of randomization to the date of death due to any cause.
Number of Participants With Clinical Laboratory Abnormalities | Time from the date of first dose of study intervention through 30-37 days after last dose of study intervention (approximately 3 years)
  laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0) and timing
Pharmacokinetics (PK): Serum concentration of PF-08634404 | Up to 37 days after the last dose of treatment
  Pre-dose and post dose concentrations of PF-08634404
Incidence of Anti-Drug Antibody (ADA) against PF-08634404 | Up to 37 days after the last dose of treatment
  To evaluate the immunogenicity of PF-08634404

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.